CLINICAL TRIAL: NCT03607188
Title: A Phase I Tolerance, Safety and Efficacy Study of Alkotinib in Patients With Advanced ALK Positive /ROS1 Positive NSCLC and Previously Treated With Chemotherapy or Crizotinib
Brief Title: Study of Alkotinib in Patients With Advanced Non Small Cell Lung Cancer
Acronym: NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZGALK001
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ZG0418 200mg QD (Experimental): ZG0418 200mg/day,oral
  Interventions: Drug: Alkotinib
- ZG0418 300mg QD (Experimental): ZG0418 300mg/day,oral
  Interventions: Drug: Alkotinib
- ZG0418 400mg QD (Experimental): ZG0418 400mg/day,oral
  Interventions: Drug: Alkotinib
- ZG0418 500mg QD (Experimental): ZG0418 500mg/day,oral
  Interventions: Drug: Alkotinib
- ZG0418 600mg QD (Experimental): ZG0418 600mg/day,oral
  Interventions: Drug: Alkotinib

INTERVENTIONS:
Drug: Alkotinib — Alkotinib 200mg QD、 Alkotinib 300mg QD、 Alkotinib 400mg QD、 Alkotinib 500mg QD、 Alkotinib 600mg QD
  Other Names: ZG0418

SUMMARY:
To explore the DLT of ZG0418 for Patients with Advanced ALK+ or ROS1+ NSCLC And Previously Treated with Chemotherapy or Crizotinib, and to determine the MTD or the R2PD.

DETAILED DESCRIPTION:
The study is a randomized, double-blind phase 1 trial including 2 sequential parts: single ascending dose(SAD) part,multiple ascending dose(MAD) part. SAD and MAD are dose-escalated tolerant study designing. The aims of the study as below:

1. Evaluating the safety and tolerance of ZG0418 in ALK+ NSCLC.
2. Evaluating the fasting pharmacokinetic parameters of ZG0418 in ALK+ NSCLCJaktinib.
3. Evaluating the postprandial pharmacokinetic parameters of ZG0418 in ALK+ NSCLC.
4. Analysis the metabolites of ZG0418

ELIGIBILITY:
Inclusion Criteria:

1. Advanced ALK+ or ROS1+ NSCLC And Previously Treated with Chemotherapy or Crizotinib
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2.
3. Life expectancy of at least 12 weeks.
4. Ability to swallow and retain oral medication.
5. Adequate organ system function, defined as follows:

   1. Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
   2. Platelets ≥75 x 10^9/L
   3. Hemoglobin ≥9 g/dL (≥90 g/L) Note that transfusions are allowed to meet the required hemoglobin level
   4. Total bilirubin ≤1.5 times the upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)

      ≤2.5 x ULN if no liver involvement or ≤5 x ULN with liver involvement.
   6. Creatinine 1.5 x ULN.
6. Brain metastases allowed if asymptomatic at study baseline.
7. Patients must have measurable disease per RECIST v. 1.1.

Exclusion Criteria:

1. chemotherapy, radiation therapy, immunotherapy within 4 weeks.
2. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of study medications.
3. uncontrolled mass of pleural effusion, pericardial effusion, and peritoneal effusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
MTD | Day1 to Day25
  Evaluating Dose-Limiting Toxicities (DLTs) from the individuals taking orally dose-escalated Alkotinib

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Doctor, Principal Investigator — Shanghai Eastern Hospital
Locations (1):
- Shanghai Eastern Hospital, Shanghai, Shanghai Municipality, China